CLINICAL TRIAL: NCT05075005
Title: A Randomized Control Trial Studying the Effects of Terrain Variation on Intrinsic Foot Musculature in Healthy Individuals and Individuals With Plantar Fasciitis:
Brief Title: The Effects of Terrain Variation on Intrinsic Foot Musculature in Healthy Individuals and Individuals With Plantar Fasciitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202100081; OCR40929 (Other: UF OnCore)
Record Dates: First submitted 2021-09-10; First posted 2021-10-12 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: A prospective, randomized control trial of patients randomly assigned to one of two groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Cohort (Active Comparator): Treatment Cohort: Will utilize a minimalist shoe (Vibram® Fivefingers) and follow the training protocol described below for training on natural terrain.
  Interventions: Other: Treatment Cohort; Other: Control Cohort
- Control Cohort (Experimental): Control Cohort: Will utilize the same minimalist shoe and follow the same training schedule as the treatment group, with the modification of training on hardscapes.
  Interventions: Other: Treatment Cohort; Other: Control Cohort

INTERVENTIONS:
Other: Treatment Cohort — Subjects will walk on a specified University of Florida Natural Area Teaching Laboratory's (NATL) nature trail for approximately 30 minutes, three times per week for 8 weeks while wearing the minimalist shoes provided by the study team. Time, distance, and GPS walking route will be recorded utilizing the MapMyRun smartphone application, which is free to download and easy to use. The study team will assist each subject with downloading the application onto their smartphone and provide a brief training on app use at their pre-trial visit. Subjects will be asked to save each training session within the app to report to the study team upon completion of the 8-week training protocol. Subjects will be instructed to walk at a comfortable pace and to stop if they begin experiencing increased pain or discomfort.
Other: Control Cohort — Subjects will walk on hardscapes (e.g. sidewalk, asphalt, track, etc) for approximately 30 minutes, three times per week for 8 weeks while wearing the minimalist shoes provided by the study team. Similarly to the treatment group, subjects will be asked to utilize the MapMyRun smartphone application to record their training sessions. Subjects will be instructed to walk at a comfortable pace and to stop if they begin experiencing increased pain or discomfort.

SUMMARY:
Modern footwear has been implicated as a contributor to foot pathology and changes in the biomechanics of gait. In addition to footwear, the investigators propose that the lack of terrain variation may directly contribute to the development of common foot pathologies, resulting from decreased intrinsic foot muscle function. This study will examine the current understanding of terrain variation on foot musculature strength and its possible correlation with structural and functional changes within the foot.

DETAILED DESCRIPTION:
The Human foot is one or the most complicated structures in the conveyance of normal gait, with its 26 bones, 33 articulations, 19 individual intrinsic muscles and direct contribution from all of the lower leg musculature. It also contains a complexity of ligamentous structures that not only act as stabilizers, but also store and release energy in a spring like fashion (Ker 1987). This group of anatomical structures is modulated by a complex system of mechanoreceptors that allow for adaptation to a multitude of varying terrain, while maintaining stability and control. (Franklin 2018) Thus the investigators see the structural, spring and muscular systems all coordinating together to allow for bipedal gait through the natural world.

Multiple observational studies have found an exceptionally low prevalence of common foot pathologies in unshod populations that ambulate on variable terrain daily (Shulman, Choi). At the same time, these same pathologies have become increasingly common in western societies. These findings suggest that something about the western lifestyle is contributing to the development of common foot pathologies. Modern footwear has already been implicated as a contributor to foot pathology and changes in the biomechanics of gait. In a study by K. D'AoÛt et al. on an unshod vs shod Indian population, they found that barefoot walkers had a more equal distribution of peak pressures over the entire load carrying surface than in the habitually shod subjects. The shod subjects had regions of very high or very low peak pressures throughout the load carrying surface.

The increase prevalence of foot pain in the developed world has long been recognized as a significant risk factor for ambulatory disability, (Hill, C. 2008) with plantar fasciitis and hallux valgus being two of the most common causes of foot discomfort presenting in the clinical setting today. Plantar fasciitis accounts for approximately 13% of all foot symptoms requiring professional medical treatment and is believed to be the result of weakening of the intrinsic foot musculature and chronic overload to the plantar foot supportive structure. (Buchanan, B. 2020). Intrinsic foot muscle function seems to play and import role in the development of foot pathology, and is one of the key factors effecting foot health.

The lack of terrain variation found in urbanized western society may directly contribute to the development of foot pathologies. Terrain variation in a minimally shod foot should allow for more coordination and strengthening of the muscular and spring like systems within the foot, through the increase and variation of stimuli encountered by its mechanoreceptors. Lack of terrain variation most probably contributes to a decreased intrinsic foot muscle function and response. There have been many studies showing the correlation between improved intrinsic foot musculature strength and the reduction of foot pain and discomfort, but to date, there are no studies that examined the relationship between terrain variation and intrinsic foot muscle function and strength.

ELIGIBILITY:
Inclusion Criteria for Group A:

* Patients presenting to the University of Florida Orthopaedics and Sports Medicine Institute with pain on the plantar medial or central heel for greater than 60 days with the following features
* Pain upon palpation, or insidious pain onset
* Pain accentuated after long periods of weight bearing activities or after periods of rest
* A reduction in pain following light activities (McPoil et al., 2008)
* Failure to respond to treatment modalities for 6 months, including plantar fascia and muscle stretching, nonsteroidal anti-inflammatory medication, supportive insoles, and night splints
* Age >18 years

Inclusion Criteria for Group B:

* Healthy individuals in the general population of Gainesville and surrounding areas
* Age >18

Exclusion Criteria for Group A:

* History of lower leg or foot surgery, hindfoot trauma or fracture of the affected limb within the previous year.
* Diagnosis of diabetic neuropathy, fibromyalgia, neurological disease, Achilles tendinopathy, metatarsalgia, tarsal tunnel syndrome or heel pad syndrome
* Body Mass Index (BMI) > 35
* Currently taking or applying any anti-inflammatory medication or medication to control nerve pathology, prescription or over the counter
* Third trimester pregnancy

Exclusion Criteria for Group B:

* Any foot or lower limb pathology resulting in discomfort or gait limitation
* Diagnosis of diabetic neuropathy, fibromyalgia, neurological disease
* BMI >35
* Currently taking or applying any anti-inflammatory medication or medication to control nerve pathology, prescription or over the counter
* Third trimester pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Revised Foot Function Index (FFI-R) | Up to 9 weeks
  34 questions rated on a scale from 1 to 4, will be used to evaluate change in overall foot function, foot health, and quality of life at trial onset, at the end of each week throughout the training protocol and upon completion of the training protocol (total of 9 times).
Visual Analog Scale (VAS) | Up to 9 weeks
  Zero millimeters on the VAS corresponds to 'no pain,' while 100 millimeters on the VAS corresponds to 'worst pain imaginable.' The participant will be asked to draw a vertical line perpendicular to the VAS line at the point that depicts their pain intensity on average throughout the week. The distance from the zero millimeter line to the participant's vertical mark will be measured to yield a score that ranges from 0 to 100. The change in these measurements is being assessed at the end of each week of the training protocol and upon completion of the training protocol (total of 9 times).

CONTACTS AND LOCATIONS:
Overall Officials: Antony Merendino, DPM, Principal Investigator — University of Florida
Locations (1):
- UF Health Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No